CLINICAL TRIAL: NCT05847946
Title: The Effect of Kinesio Taping on Pain and Disability in Pregnancy-Related Low Back Pain: A Randomized Clinical Study
Brief Title: The Effect of Kinesio Taping on Pain and Disability in Pregnancy-Related Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Collaborators: HASAN GERÇEK (Unknown); ŞERİFE İREM DÖNER (Unknown); BAYRAM SÖNMEZ ÜNÜVAR (Unknown)
Responsible Party: Principal Investigator, Hafize Dağ Tüzmen, LECTURER, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kinesio
Record Dates: First submitted 2023-04-18; First posted 2023-05-08 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Pregnancy-related Low Back Pain
Keywords: Pregnancy; Low back pain; Function; Kinesiologic tape; core stabilization
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Core stability and pelvic floor exercises will be compared with kinesiotape application.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotape application (Experimental): In addition to core stabilization and pelvic floor exercises, kinesiotape will be applied to the paraspinal muscles in the lumbar region 2 times a week for a total of 8 times.
  Interventions: Other: Kinesio tape application and Core stabilization home program
- Core stability and pelvic floor exercises group (Active Comparator): Participants will perform core stabilization and pelvic floor exercises 5 days a week for 4 weeks.
  Interventions: Other: Core stabilization home program

INTERVENTIONS:
Other: Kinesio tape application and Core stabilization home program — Participants in the kinesiotape group will receive 2 sessions of kinesiotape per week, in addition to the core stabilization home program, 5 days a week for 4 weeks.
  Arms: Kinesiotape application
Other: Core stabilization home program — Core stabilization exercises will be given to the participants as a home exercise program.
  Arms: Core stability and pelvic floor exercises group

SUMMARY:
Pregnant women may experience pregnancy-related low back pain and this pain may negatively affect function. There are studies in the literature that Kinesiotape applications improve pain. There is no study examining the effect of Kinesiotape application in addition to exercise on pregnancy-related low back pain and function. At the end of our study, we will compare the effects of Kinesiotape application for a total of 8 sessions for 4 weeks on pain and function.

DETAILED DESCRIPTION:
Kinesio tape (KT) application is a physiotherapy method whose use has increased in recent years in the treatment of chronic pain. Kinesio tape, an alternative method to support fascia, muscles and joints, Dr. Developed by Kenzo Kase. Although the therapeutic effects of the KT method are still unclear, the putative therapeutic effects include facilitating muscle activity, providing sensory stimuli to the skin, muscles or facial structures, and regulating joint range of motion (ROM) . KT method increases blood and lymph circulation by lifting the skin, and prevents pain by reducing nociceptive stimuli . KT has been administered to pregnancy to improve low back pain. In addition to publications showing that KT can reduce pregnancy-related low back pain, there are studies showing that it has no effect compared to the control group . The aim of this study is to examine the effect of 8 sessions of KT applied in addition to 4-week core stabilization exercises on pain and quality of life in pregnant women with pregnancy-related low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age between 18 and 40 years, any birth,
* gestational age between 13 and 30 weeks,
* low back pain anywhere from T12 to gluteal fold without leg pain and at least moderate pain intensity (VAS ≥ 4).

Exclusion Criteria:

* Known or suspected orthopedic or rheumatological disorders such as scoliosis,
* spinal injuries,
* ankylosing spondylitis or rheumatoid arthritis;
* intervertebral disc pathology;
* a history of low back pain before pregnancy;
* twin pregnancy or fetal anomaly; and any uncontrolled medical conditions

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women will be included in the study.
Enrollment: 42 (Actual)
Dates: Start 2023-06-04 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline pregnancy-related low back Pain at 4 weeks | Baseline and after 4 weeks intervention
  Pain will be assessed with a 10 cm visual analog scale at night, at rest and during activity. "0" means no pain and "10" means unbearable pain. The assessment will be done before and at the end of the study.
Change from Baseline Function at 4 weeks | Baseline and after 4 weeks intervention
  Function will be assessed with the Oswestry Low Back Pain Disability Questionnaire. The higher the score on the scale, the greater the loss of function. Assessment will be done before and at the end of the study.

SECONDARY OUTCOMES:
Change from Baseline Health Quality at 4 weeks | Baseline and after 4 weeks interventionBaseline and after 4 weeks intervention
  Quality of life will be assessed with the Short Form 36. The higher the score on the scale, the better the quality of life. The assessment will be done before and at the end of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No